CLINICAL TRIAL: NCT04065269
Title: ATARI: ATr Inhibitor in Combination With Olaparib/Durvalumab (MEDI4736) in Gynaecological Cancers With ARId1A Loss or no Loss
Brief Title: ATr Inhibitor in Combination With Olaparib/Durvalumab (MEDI4736) in Gynaecological Cancers With ARId1A Loss or no Loss
Acronym: ATARI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICR-CTSU/2018/10066; 2018-003779-36 (EudraCT Number)
Record Dates: First submitted 2019-08-01; First posted 2019-08-22 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Gynaecological Cancers
Keywords: Clear cell ovarian carcinoma; Clear cell endometrial carcinoma; Endometrioid carcinoma; Carcinosarcoma; Cervical carcinoma; ARID1A; Endometrial cancer
MeSH Terms: conditions — Carcinoma, Endometrioid; Carcinosarcoma; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — ceralasertib; olaparib; durvalumab

STUDY DESIGN:
Intervention Model Description: Open-label, multiple two-stage parallel cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1A: ceralasertib (AZD6738) (Experimental): Women with relapsed ovarian (fallopian tube / primary peritoneal) and endometrial (uterus) clear cell carcinomas with loss of ARID1A expression treated with single agent AZD6738.
  Interventions: Drug: Ceralasertib
- 1B: ceralasertib (AZD6738) + olaparib (Experimental): In second stage of trial, opening of this cohort depends on response rate in cohort 1A during first stage of trial.
  Women with relapsed ovarian (fallopian tube / primary peritoneal) and endometrial (uterus) clear cell carcinomas with loss of ARID1A expression treated with AZD6738 in combination with olaparib.
  Interventions: Drug: Ceralasertib; Drug: Olaparib
- 2: ceralasertib (AZD6738) + olaparib (Experimental): Women with relapsed ovarian (fallopian tube / primary peritoneal) and endometrial (uterus) clear cell carcinomas with NO loss of ARID1A expression treated with AZD6738 in combination with olaparib.
  Interventions: Drug: Ceralasertib; Drug: Olaparib
- 3: ceralasertib (AZD6738) + olaparib (Experimental): Women with other rare relapsed gynaecological cancers (endometrioid ovarian carcinoma, endometrioid endometrial carcinoma, cervical adenocarcinoma, cervical squamous, ovarian carcinosarcoma and endometrial carcinosarcoma) irrespective of ARID1A status, treated with AZD6738 in combination with olaparib.
  Interventions: Drug: Ceralasertib; Drug: Olaparib
- 4: ceralasertib (AZD6738) + durvalumab (Experimental): Women with endometrial cancers (serous, clear cell, endometroid, carcinosarcoma) with ARID1A loss.
  Interventions: Drug: Ceralasertib; Drug: Durvalumab
- 5: ceralasertib (AZD6738) + durvalumab (Experimental): Women with endometrial cancers (serous, clear cell, endometroid, carcinosarcoma) with NO loss of ARID1A.
  Interventions: Drug: Ceralasertib; Drug: Durvalumab

INTERVENTIONS:
Drug: Ceralasertib — ATR inhibitor
  Other Names: AZD6738
Drug: Olaparib — PARP inhibitor
  Arms: 1B: ceralasertib (AZD6738) + olaparib; 2: ceralasertib (AZD6738) + olaparib; 3: ceralasertib (AZD6738) + olaparib
Drug: Durvalumab — Anti-PD-L1 immunotherapy
  Other Names: MEDI4736
  Arms: 4: ceralasertib (AZD6738) + durvalumab; 5: ceralasertib (AZD6738) + durvalumab

SUMMARY:
ATARI trial tests the ATR inhibitor drug ceralasertib (AZD6738) alone and in combination with either a PARP inhibitor drug called olaparib, or an anti-PD-L1 immunotherapy called durvalumab (MEDI4736) in patients with relapsed gynaecological cancers to assess the response in groups of patients selected based on their cancer cell subtype and the presence of an abnormality in the ARID1A gene.

DETAILED DESCRIPTION:
ATARI is a multi-centre, open-label, multiple two-stage parallel cohorts phase II clinical trial for patients with relapsed gynaecological cancers, with ARID1A-deficient ('loss') and "no loss."

The trial tests the ATR inhibitor drug ceralasertib (AZD6738) alone and in combination with either a PARP inhibitor drug called olaparib, or an anti-PD-L1 immunotherapy called durvalumab (MEDI4736) to assess the response in groups of patients selected based on their cancer cell subtype and the presence of an abnormality in ARID1A.

The treatment groups are: 1A - Women with clear cell subtype with (ovarian/uterus) ARID1A loss treated with ceralasertib. 1B - Women with clear cell subtype with (ovarian/uterus) ARID1A loss treated with ceralasertib and olaparib. 2 - Women with clear cell subtype (ovarian/uterus) with no ARID1A loss treated with AZD6738 and olaparib. 3 - Women with other rare gynaecological cancers (carcinosarcoma, cervical, endometrioid type) irrespective of ARID1A loss treated with ceralasertib and olaparib. 4 - Women with endometrial cancers (serous, clear cell, endometroid, carcinosarcoma) with ARID1A loss treated with ceralasertib and durvalumab. 5 - Women with endometrial cancers (serous, clear cell, endometroid, carcinosarcoma) with no ARID1A loss treated with ceralasertib and durvalumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed progressive or recurrent gynaecological carcinomas of the following histological subtypes:

   Cohorts 1A, 1B, 2 and 3:
   * Clear cell (Ovarian, endometrial or endometriosis-related, (>50% clear cell carcinoma with no serious differentiation)
   * Endometrioid (ovarian, endometrial or endometriosis-related)
   * Cervical (adenocarcinomas or squamous)
   * Carcinosarcomas (ovarian or endometrial)

   Cohorts 4 and 5:

   • Endometrial carcinomas (serous, clear cell, endometrioid, carcinosarcoma) Note: patients who have an original diagnosis based on cytology only will not be eligible for entry into the study unless a biopsy confirming above histology is performed
2. Histological tissue specimen (tissue block or 8-10 unstained slides) must be available (specimen can be the sample at diagnosis or taken at relapse). Otherwise, a biopsy must be carried out to obtain sufficient tissue for histological assessment
3. Evidence of radiological disease progression since last systemic anti-cancer therapy and prior to trial entry
4. Patients who have progressed after ≥1 prior platinum containing regimen. Platinum-based therapy does not need to be the last treatment prior to study entry. For Cohorts 1A, 1B, 2 and 3, patients who have disease progression within 6 months of last dose of a platinum-containing regimen, no more than two further lines of systemic therapy are permitted prior to trial entry
5. Patients entering Cohorts 4 or 5 must have had prior anti-PD-1/anti-PD-L1/anti-CTLA-4 immunotherapy treatment, with a minimum duration of treatment is 6 weeks. Other previous immunotherapy treatments may be permissible following discussion with the Chief Investigator and ICR-CTSU. Patients who experienced toxicity leading to permanent discontinuation of prior immunotherapy are ineligible.

   * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
   * Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enrol if they are stably maintained on appropriate replacement therapy and are asymptomatic.
   * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
6. Body weight >30kg (Cohorts 4 and 5 only)
7. Measurable disease by RECIST criteria v1.1, which can be accurately assessed at baseline by CT (or MRI where CT is contradicted or unclear). Patients with CA125 progression in the absence of measurable disease will NOT be eligible
8. ECOG performance status 0 or 1 with no deterioration over the previous 2 weeks
9. Life expectancy > 16 weeks
10. Adequate hepatic, bone marrow, coagulation and renal function as defined by the following values within 14 days prior to starting treatment:

    All cohorts:
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
    * Platelet count ≥ 100 x 109/L with no platelet transfusion in the past 28 days
    * Total bilirubin ≤1.5 x ULN (where bilirubin rise > 1.5 x ULN due to Gilbert's syndrome a conjugated bilirubin ≤1.5 x ULN is required)
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤2.5 x ULN if no demonstrable liver metastases or ≤5 times ULN if patient has documented liver metastases

    Cohort 1A, Cohort 4 and Cohort 5:
    * Haemoglobin ≥9.0 g/dL with no blood transfusion in the past 14 days
    * Glomerular filtration rate (GFR) ≥45 mL/min (estimated using Cockcroft-Gault equation, MDRD, 24hr urine collection as appropriate)

    Cohort 1B, Cohort 2 and Cohort 3:
    * Haemoglobin ≥10.0 g/dL with no blood transfusion in the past 14 days
    * Glomerular filtration rate ≥51 mL/min (estimated using Cockcroft-Gault equation, MDRD, 24hr urine collection as appropriate)
11. No significant medical illness which in the opinion of the Investigator would preclude entry to ATARI
12. Women of child-bearing potential who are confirmed NOT to be pregnant. This should be evidenced by a negative urine or serum pregnancy test within 72 hours prior to start of trial treatment (cohort 4 and 5 must be serum at screening). Patients will be considered to be not of child-bearing potential if they are:

    * Post-menopausal - defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments, OR women under 50 years old who have been amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments and have serum follicle-stimulating hormone (FSH), luteinizing hormone (LH) and plasma oestradiol levels in the post-menopausal range for the institution
    * Able to provide documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
    * Radiation or chemotherapy-induced oophorectomy or menopause with > 1 year since last menses
13. Patients with prior synchronous tumours or history of prior malignancy are eligible provided there is biopsy evidence that the disease measurable on CT and/or MRI is of the histological subtypes stated in 1
14. Willingness to commit to scheduled visits, treatments plans, laboratory tests and study procedures
15. Able to swallow, absorb, retain oral medication
16. Able to provide written, informed consent Exclusion Criteria
17. Patients receiving, or having received

    * Cohort 1A, Cohort 4 and Cohort 5: Prior treatment with ATR inhibitor
    * Cohort 1B, Cohort 2 and Cohort 3: Prior treatment with ATR or PARP inhibitors
18. Patients receiving, or having received:

    * cytotoxic treatment for their malignancy within 21 days prior to Cycle 1 Day 1
    * exposure to a small molecule IP within 30 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1. The minimum washout for immunotherapy is 42 days
    * treatment with bevacizumab within 30 days prior to Cycle 1 Day 1
    * palliative radiotherapy within 21 days prior to Cycle 1 Day 1 (with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study treatment). Patients can receive bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to commencing study treatment.
19. Treatment with any other investigational medicinal product within the 4 weeks prior to trial entry
20. Receiving, or having received, concomitant medications, herbal supplements and/or foods that are strong or moderate inhibitors or inducers of CYP3A4 and/or CYP1A2 for cohorts 1B, 2 and 3, and strong inhibitors or inducers of CYP3A4 and/or CYP1A2 for cohorts 1A, 4 and 5, sensitive CYP3A4 and/or CYP1A2 substrates or CYP3A4 and/or CYP1A2 substrates with a narrow therapeutic index that significantly modulate CYP3A4 and/or CYP1A2 or P-gp activity (washout period 5 half-lives or three weeks for St. John's Wort). Note these include common azole antifungals, macrolide antibiotics and other medications (Refer to Sections 22, 23 & 24 and Appendix A6 for further details)
21. Pregnant or lactating women.
22. Women of childbearing age and potential who are not willing to use one highly effective form of contraception AND a condom as detailed in Section 5.5.1
23. Any other malignancy which has been active or treated within the past three years, with the exception of cervical intra-epithelial neoplasia and non-melanoma skin cancer
24. Clinical/radiological evidence of bowel obstruction (e.g. hospitalisation) or symptoms of sub-acute bowel obstruction within 6 weeks prior to trial entry
25. Any clinically significant haematuria (as deemed by the investigator)
26. With the exception of alopecia, any unresolved toxicities from prior therapy should be no greater than CTCAE Grade 2 at trial entry
27. Clinically significant cardiac disease currently or within the last 6 months including:

    a. Pre-existing arrhythmia: i. Mean resting QTc >470 msec obtained from 3 electrocardiograms (ECGs) performed 2-5 minutes apart at study screening (within 14 days prior to Cycle 1 Day 1) using the Fredericia formula ii. Clinically important abnormalities in rhythm, conduction or morphology of resting ECG (including complete left bundle-branch block, third degree heart block) b. Any factor increasing the risk of QTc prolongation or arrhythmia, including: i. Hypokalaemia ii. Congenital long QT syndrome iii. Immediate family history of long QT syndrome or unexplained sudden death below the age of 40 years c. Unstable angina pectoris d. Acute myocardial infarction e. Unstable cardiac arrhythmias f. Cardiac failure i. Known reduced LVEF <55% ii. New York Heart Association (NYHA) class II, III or IV cardiac failure g. Uncontrolled hypertension (≥ grade 2) requiring clinical intervention (Cohort 4 and Cohort 5 only)
28. Clinically relevant orthostatic hypotension
29. Patients who have a diagnosis of ataxia telangiectasia
30. Major surgery within 4 weeks prior to starting trial drug (excluding placement of vascular access) or minor surgery (excluding tumour biopsies) within 2 weeks of starting trial.Local surgery of isolated lesions for palliative intent is acceptable
31. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
32. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
33. Known leptomeningeal involvement or brain metastases, unless asymptomatic, treated (with no evidence of progression since completion of CNS-directed therapy), presence of disease outside the CNS and stable off steroids for at least 4 weeks prior to registration
34. Known hypersensitivity to investigational drugs or excipients
35. Receiving, or having received during the four weeks prior to starting trial drug, corticosteroids at a dose >10mg prednisolone/day or equivalent for any reason
36. Any haemopoietic growth factors (e.g., G-CSF, GM-CSF) and blood transfusions within 14 days prior to trial entry. Use of erytropoeitin is not permitted for 4 weeks prior to Cycle 1 Day 1 and for the duration of the study
37. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases that places the patient at unacceptable risk of toxicity or non-compliance e.g., severe hepatic impairment, extensive interstitial lung disease on high resolution CT scan (bilateral, diffuse, parenchymal lung disease), uncontrolled chronic renal diseases (glomerulonephritis, nephritic syndrome, Fanconi Syndrome or Renal tubular acidosis), current unstable or uncompensated respiratory or cardiac conditions, active bleeding diatheses or active infection including hepatitis B, hepatitis C, and immunocompromised patients e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV). Screening for chronic conditions is not required
38. Judgment by the Investigator that the patient is unsuitable to participate in the study and/or the patient is unlikely to comply with study procedures, restrictions and requirements
39. Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of study drug
40. Patients with uncontrolled seizures
41. Active infection requiring systemic antibiotics, antifungal or antiviral drugs
42. Patients with myelodysplastic syndromes (MDS)/acute myeloid leukaemia (AML), or with features suggestive of MDS/AML
43. Concurrent severe and/or uncontrolled medical condition (e.g., severe COPD, severe Parkinson's disease, active inflammatory bowel disease) or psychiatric condition (e.g. psychiatric disorder prohibiting obtaining informed consent)
44. Any contraindication to the combination anti-cancer agent (ceralasertib/olaparib or ceralasertib/durvalumab) as per local prescribing information
45. Patients unable to swallow orally administered medication
46. Patients in receipt of any live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study treatment. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study drug and up to 30 days after the last dose of study drug.
47. Patients with a confirmed COVID-19 infection by PCR test who have not made a full recovery

    In addition to the above and specific for Cohorts 4 and 5 only:
48. Any concurrent chemotherapy, IP, biological, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
49. Persisting (>4 weeks) severe pancytopenia due to previous therapy rather than disease (ANC <0.5 x 109/L or platelets <50 x 109/L)
50. History of organ transplant that requires use of immunosuppressive medications including, but not limited to systemic corticosteroids at doses >10mg/day of prednisone or equivalent, methotrexate, azathioprine and tumour necrosis factor alpha (TNF-α) blockers. Use of immunosuppressive medications for the management of IMP-related AEs is acceptable
51. Active or prior documented autoimmune or inflammatory disease within the past 3 years (including, but not limited to inflammatory bowel disease [e.g., Crohn's disease or colitis], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, Wegener syndrome, Hashimoto syndrome, hyperthyroidism, Sjogren's syndrome, glomerulonephritis, multiple sclerosis, vasculitis, rheumatoid arthritis, idiopathic pulmonary fibrosis, pneumonitis, organising pneumonitis, hepatitis, sarcoidosis, active tuberculosis.

The following are exceptions to this criterion:

* Patients with vitiligo or alopecia, patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement. Any chronic skin condition that does not require systemic therapy, patients without active disease in the last 5 years may be included but only after consultation with the ATARI Chief Investigator. Patients with celiac disease controlled by diet alone.

  52. History of another primary malignancy except for:
* Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of the study drug and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease 53. History of active primary immunodeficiency 54. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of durvalumab. The following are exceptions to this criterion:
* Intranasal, inhaled, topical steroids or local steroid injections (e.g., intra articular injection)
* Systemic corticoids at physiologic doses not to exceed 10mg/day of predisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan medication)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Confirmed overall objective response rate (complete or partial response) as defined by RECIST version 1.1. | From start of treatment until treatment discontinuation - minimum follow-up of 16 weeks (if not progressed earlier), up to max study period (estimated 36 months).
  A patient will be said to have had an overall objective response if they have a complete/partial response as assessed radiologically according to RECIST 1.1 at any point during trial treatment. A second scan to confirm response will be taken ≥ 4 weeks after the first scan showing an objective response.

SECONDARY OUTCOMES:
Disease control rate | From start of treatment until treatment discontinuation - minimum follow-up of 16 weeks (if not progressed earlier), up to max study period (estimated 36 months).
  The proportion of patients experiencing complete or partial response, or stable disease lasting at least 16 weeks from start of treatment as assessed radiologically by RECIST version 1.1.
Duration of disease control | From start of treatment until treatment discontinuation - minimum follow-up of 16 weeks (if not progressed earlier), up to max study period (estimated 36 months).
  Length of maintained response, measured according to RECIST v1.1
Progression Free Survival (PFS) | From start of treatment until progression or death, whatever occurs first - estimated 6-9 months, up to max study period (36 months).
  Measured according to RECIST v1.1 or death. Time to last tumour assessment will be used if patient has not progressed or died, and PFS time for the patient will be considered censored. PFS will be used to calculate the proportion of patients alive and free of progression at 6 months.
Time to Progression (TTP) | From start of treatment until disease progression - estimated 6-9 months, up to max study period (36 months)
  Measured according to RECIST v 1.1 or clinical progression of disease. Time to last tumour assessment will be used if patient has not progressed, and the patient will be considered censored. If the patient has died without prior progression, the patient will be censored at the date of death. Death will not count as a TTP event.
Proportion of patients experiencing drug interruption, reduction or discontinuation due to drug related adverse events | Assessed throughout the treatment period, up to and including the 30-day follow-up period - estimated 7 months, up to max study period (36 months).
  Adverse events thought to be related to drug will be graded according to NCI-CTCAE version 5.0, and coded using MedDRA (current version). Any dose reductions and delays in administration of drug due to toxicity will also be collected.
Overall Survival (OS) | From start of treatment until death - estimated 9 months, up to max study period (36 months).
  Defined by the time from start of treatment until death

CONTACTS AND LOCATIONS:
Overall Officials: Susana Banerjee, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (9):
- Canada (3):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - University of Montreal Hospital Centre, Montreal, Quebec
- United Kingdom (6):
  - Royal United Hospital, Bath
  - Western General Hospital, Edinburgh
  - The Beatson, Glasgow
  - The Royal Marsden NHS Foundation Trust, London
  - Imperial College NHS Trust, London
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith G, Alholm Z, Coleman RL, Monk BJ. DNA Damage Repair Inhibitors-Combination Therapies. Cancer J. 2021 Nov-Dec 01;27(6):501-505. doi: 10.1097/PPO.0000000000000561. PMID 34904813